CLINICAL TRIAL: NCT01538745
Title: Low Dose Ketamine (LDK) Versus Morphine for Acute Pain Control in the Emergency Department
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Brooke Army Medical Center (U.S. Federal Agency)
Collaborators: U.S. Air Force Office of the Surgeon General (U.S. Federal Agency)
Responsible Party: Principal Investigator, Joshua Miller, Joshua Miller, Maj, USAF, MC, Brooke Army Medical Center
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: C.2011.173
Record Dates: First submitted 2012-02-21; First posted 2012-02-24 (Estimated); Results first posted 2021-02-04 (Actual); Last update posted 2021-02-04 (Actual); Status verified 2021-02

CONDITIONS: Abdomen, Acute; Other Acute Pain; Flank Pain; Back Pain; Musculoskeletal Pain
Keywords: Pain; Emergency Department; Morphine; Ketamine
MeSH Terms: conditions — Abdomen, Acute; Flank Pain; Back Pain; Musculoskeletal Pain; Pain; Emergencies | interventions — Ketamine; Morphine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Ketamine (Experimental): 0.3 MG/KG IV KETAMINE ADMINISTERED OVER 5 MINUTES. MAX DOSE OF 25MG.
  Interventions: Drug: Ketamine
- Morphine (Active Comparator): 0.1 MG/KG IV MORPHINE ADMINSITERED OVER 5 MINUTES. MAX DOSE 8MG.
  Interventions: Drug: Morphine

INTERVENTIONS:
Drug: Ketamine — 0.3 mg/kg ketamine Intravenous push (IVP) over 5 minutes. Total of two possible doses.
  Other Names: Ketalar
  Arms: Ketamine
Drug: Morphine — 0.1 mg/kg Morphine IVP over 5 minutes. Total of two possible doses.
  Other Names: MS Contin; Roxanol; Kadian; Avinza
  Arms: Morphine

SUMMARY:
The purpose of this study is to compare the safety and effectiveness of intravenous low dose ketamine (LDK) to the industry standard of morphine (MOR) in regards to controlling acute pain in the emergency department.

Both LDK and morphine have side effects. The amount and character of these side effects will be compared. Additionally, the degree of sedation or agitation will be specifically measured. The aim of this current study is to make this comparison and shift the evidence for LDK use from the anecdotal to the scientific.

DETAILED DESCRIPTION:
Phase 1 is a randomized, controlled, double-blinded study comparing the use of low-dose ketamine (LDK) to morphine for acute pain control in emergency department patients. A convenience sample of subjects will be enrolled from a population of patients aged 18-50 who present to the Brooke Army Medical Center Emergency Department with acute abdominal pain, flank/lumbar back pain and/or pain to the extremities. To take part in the study, a need for opioid analgesia must be indicated by the treating physician in addition to the patient meeting all other study criteria.

The patient will then be randomized into one of the two treatment arms. Prior to receiving either the study medication (ketamine) or the active control (morphine) the patient will be asked to rate their pain on a numeric rating scale (NRS) with 0 being no pain and 10 being the worst pain possible. Their baseline vital signs (blood pressure, heart rate, respiratory rate and oxygen saturation) will also be documented. These vital signs and the NRS will be reassessed at 5, 10 and 20 minutes post medication dosage. At 20 minutes they will also document a Richmond Agitation Sedation Scale (RASS) score and will ask the patient if they require additional pain medication. If the patient denies the need for a second dose of medication they will continue to be re-assessed every 20 minutes (vital signs, NRS, and RASS) until either inpatient admission, discharge home, transfer to the operating room or until a total of 120 minutes after initial dosing.

If at any time during the study the patient requires a second dose of pain medication, following the administration of the med, they will be assessed for vital signs at 5,10 and 20 minutes after the dose. At 20 minutes, a RASS score and NRS score will also be documented. They will then be re-assessed every 20 minutes (vital signs, NRS, and RASS) until either inpatient admission, discharge home, transfer to the operating room or until a total of 120 minutes after initial dosing.

If they require a third dose of pain medication at any time during the study, this is considered a treatment failure and the treating physician will be contacted to provide any further pain control.

The second phase of the study will be observational. An anonymous satisfaction survey will be provided to the treating nurse, physician or physicians assistant (PA) of the patients recruited from part one of the study. The purpose of conducting the survey is so that an observation point of view can be added to the data to provide a measure of how well the patient's pain was controlled.

ELIGIBILITY:
Inclusion Criteria:

* Patients age 18-59 who present to the Brooke Army Medical Center Emergency Department with acute (less than 10 days) abdominal pain, flank/lumbar back pain and or/pain to the extremities, and of sufficient severity in the judgement of the ED treating physician or PA to warrant use of intravenous opioids

Exclusion Criteria:

* Poor vital sign stability hypoxia: Sats<95% hypotension: SBP<90 hypertension: SBP>180 heart rate: <50 or >120 respiratory rate: <10 or >30
* Altered mental status or intoxication
* Patient is unwilling to participate or provide informed consent
* History of chronic pain or pain syndrome with concurrent opioid medication use
* fibromyalgia
* Patient has received opioids and/or tramadol in the past 4 hours
* Prescription pain medication use (to exclude muscle relaxants, acetaminophen or NSAIDs including toradol) in the past 4 hours
* Allergy to morphine or ketamine
* Sole provider status
* Adverse reaction to morphine or ketamine in the past
* Patients, who in the opinion of the triage nurse, require immediate analgesic relief
* Patient is female of child-bearing age and unable to provide urine or serum for HCG analysis in triage
* Pregnancy or breast feeding
* Presence of oxygen dependent pulmonary disease, liver cirrhosis or Renal disease requiring dialysis. (as assessed by electronic chart review)
* Presence of Ischemic heart disease, heart failure or unstable dysrhythmias (as assessed by electronic chart review)
* Presence of intracranial mass or vascular lesion.
* Presence of psychosis or hallucinations
* Weight greater than 115kg or less than 45 kg
* History of acute ocular/head trauma
* History of increased intracranial pressure/hypertensive hydrocephalus
* Non-English speaking patients

Ages: 18 Years to 59 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 45 (Actual)
Dates: Start 2012-02; Primary Completion 2013-03 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Joshua P Miller, MD, Principal Investigator — United States Air Force
Locations (1):
- Brooke Army Medical Center, San Antonio, Texas, United States

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study took place at a Level 1 trauma center. The patient population at SAMMC consists of active duty military personnel and their family members, retirees, as well as civilians. There are approximately 75,000 visits to the SAMMC ED annually. Enrollment occurred from February 2012 to March 2013.
Pre-assignment Details: Patients were excluded if: O2 saturation <95%, SBP < 90mmHg or > 180mmHg, HR< 50 or > 120 beats per minute, RR < 10 or > 30 per minute, altered mental status, intoxication, history fibromyalgia, ischemic heart disease, heart failure or unstable dysrhythmias, required pain medication immediately and cannot wait to consent
Groups:
- Ketamine: 0.3 MG/KG IV KETAMINE ADMINISTERED OVER 5 MINUTES. MAX DOSE OF 25MG.
  Ketamine : 0.3 mg/kg ketamine IVP over 5 minutes. Total of two possible doses.
- Morphine: 0.1 MG/KG IV MORPHINE ADMINSITERED OVER 5 MINUTES. MAX DOSE 8MG.
  Morphine : 0.1 mg/kg Morphine IVP over 5 minutes. Total of two possible doses.
Period: Overall Study
Arm/Group | Ketamine | Morphine
Started | 24 | 21
Completed | 24 | 21
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Ketamine | Morphine | Total
Number analyzed (Participants) | 24 | 21 | 45
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 24 | 21 | 45
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.75 (11.87) | 29.29 (9.78) | 30.07 (10.84)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 10 | 12 | 22
  Male | 14 | 9 | 23
Region of Enrollment [Number; unit: participants]
  United States | 24 | 21 | 45

OUTCOME MEASURES:

1. Primary Outcome: Maximal Change in Numerical Rating Scale (NRS) Pain Score From Baseline NRS Pain Score
Description: Numerical Rating Scale (NRS) pain score is an 11-point rating scale for pain. With 0 being no pain and 10 being the worst pain imaginable.
Time Frame: 5,10,20,40,60,80,100,120 minutes post dose
Measure: Mean (95% Confidence Interval); unit: NRS pain scale score
Units Other Than Participants: units on a scale
Arm/Group | Ketamine | Morphine
Number analyzed (Participants) | 24 | 21
Number analyzed (units on a scale) | 11 | 11
NRS pain scale score | -4.9 [-5.75 to -4] | -5 [-7.1 to -2.9]

2. Secondary Outcome: Time to Change in NRS Pain Score
Description: Following dosage with study medication, the amount of time taken to demonstrate a change in the patient's NRS pain score. Time to Change in NRS Pain Score for the Reporting Group as a whole will be made
Time Frame: 5,10, 20,40,60,80,100,120 minutes
Measure: Mean (Standard Deviation); unit: minutes
Arm/Group | Ketamine | Morphine
Number analyzed (Participants) | 24 | 21
minutes | 5 (2.63) | 5 (2.48)

3. Secondary Outcome: Time to Maximal Change in NRS Pain Score
Description: Following dosage with study medication, the interval time taken to demonstrate the maximal change in the patient's NRS pain score will be reported for each group.
Time Frame: 5, 10, 20 minutes and then every 20 minutes to a total of 120 minutes
Measure: Median (Standard Deviation); unit: minutes
Arm/Group | Ketamine | Morphine
Number analyzed (Participants) | 24 | 21
minutes | 5 (1.7) | 120 (22.2)

4. Secondary Outcome: Incidence of Treatment Failure
Description: Requiring more than two doses of the study medication provided for adequate pain control
Time Frame: 120 minutes
Measure: Number; unit: Percentage of patients
Arm/Group | Ketamine | Morphine
Number analyzed (Participants) | 24 | 21
Percentage of patients | 25 | 14

5. Secondary Outcome: Incidence of Side Effects, Including Outlying Vital Signs
Description: The patient will be assessed for vital signs (blood pressure, heart rate, respiratory rate, oxygen saturation), and all side effects at 5,10,20 minutes following medication administration and then every 20 minutes until a total of 120 minutes from the first dose of study medication. All side effects and outlying vital signs will be documented.
Time Frame: 5,10,20,40,60,80,100,120 minutes
Measure: Number; unit: Percentage of patients
Arm/Group | Ketamine | Morphine
Number analyzed (Participants) | 24 | 21
Percentage of patients | 58 | 57

6. Secondary Outcome: Maximum Deviation From 0 on the Richmond Agitation Sedation Scale (RASS)
Description: Using 0 as the "normal/baseline" on the RASS, maximal deviation in either direction will be used to demonstrate the effect of the study medications on levels of sedation or agitation. Results will be reported as
  Richmond Agitation Sedation Scale (RASS) scores range from:
  * 4 Combative: Overtly combative, violent, immediate danger to staff
  * 3 Very agitated: Pulls or removes tube(s) or catheter(s); aggressive
  * 2 Agitated: Frequent non-purposeful movement
  * 1 Restless: Anxious but movements not aggressive. vigorous 0 Alert and calm
    * 1 Drowsy: Not fully alert, but has sustained awakening (eye-opening/eye contact) to voice (>10 seconds)
    * 2 Light sedation: Briefly awakens with eye contact to voice (<10 seconds)
    * 3 Moderate sedation: Movement or eye opening to voice (but no eye contact)
    * 4 Deep sedation: No response to voice, but movement or eye opening to physical stimulation
    * 5 Unarousable: No response to voice or physical stimulation
Time Frame: 5,10,20,40,60,80,100,120 minutes
Measure: Mean (Full Range); unit: units on a scale
Arm/Group | Ketamine | Morphine
Number analyzed (Participants) | 24 | 21
units on a scale | 0 [-3 to 3] | 0 [-2 to 1]

ADVERSE EVENTS:
Arm/Group | Ketamine | Morphine
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/21
Other Adverse Events (participants affected / at risk) | 0/24 | 0/21

LIMITATIONS AND CAVEATS:
The side effect profile associated with ketamine and morphine are different without significant overlap thus making blinding difficult.

The exclusion criteria of our study made enrollment difficult and our sample size smaller than anticipated.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes